CLINICAL TRIAL: NCT01735487
Title: Electronic Cigarette and Cognitive Functioning: (CogEcig)
Brief Title: CogEcig: Cognitive Functioning and Electronic Cigarette
Acronym: CogEcig
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita degli Studi di Catania (Other)
Responsible Party: Principal Investigator, Riccardo Polosa, Professor, Universita degli Studi di Catania
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: CogEcig
Record Dates: First submitted 2012-11-23; First posted 2012-11-28 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Tobacco Abuse Smoke
MeSH Terms: interventions — Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Own Brand cigarette (Active Comparator): Smoke Own Brand cigarette, 15 puff of cigarette.
  Interventions: Other: one high 2,4% nicotine; Other: original 7,4 mg nicotine; Other: nicotine free; Other: Ego 9mg
- One High 2,4% nicotine (Experimental): Smoke electronic cigarette One High 2,4% nicotine for a day, 15 puff of e-cigarette.
  Interventions: Other: Own Brand cigarette; Other: original 7,4 mg nicotine; Other: nicotine free; Other: Ego 9mg
- Original 7,4 mg nicotine (Experimental): Smoke electronic cigarette Original 7,4 mg nicotine for a day. 15 puff of e-cigarette.
  Interventions: Other: Own Brand cigarette; Other: one high 2,4% nicotine; Other: nicotine free
- Nicotine Free (Placebo Comparator): Smoke electronic cigarette nicotine free (15 puff)
  Interventions: Other: Own Brand cigarette; Other: one high 2,4% nicotine; Other: original 7,4 mg nicotine; Other: Ego 9mg
- EGO 9mg (Experimental): Smoke electronic cigarette EGO for a day (15 puff)
  Interventions: Other: Own Brand cigarette; Other: one high 2,4% nicotine; Other: original 7,4 mg nicotine; Other: nicotine free

INTERVENTIONS:
Other: Own Brand cigarette — Smoke, 15 puff of, Own Brand cigarettes;
  Arms: EGO 9mg; Nicotine Free; One High 2,4% nicotine; Original 7,4 mg nicotine
Other: one high 2,4% nicotine — Smoke, 25 puff, of electronic cigarette one high 2,4% nicotine
  Other Names: Categoria electronic cigarette one high 2,4% nicotine
  Arms: EGO 9mg; Nicotine Free; Original 7,4 mg nicotine; Own Brand cigarette
Other: original 7,4 mg nicotine — Smoke, 15 puff, of Categoria electronic cigarette 7,4 mg nicotine
  Other Names: Categoria electronic cigarette 7,4 mg nicotine
  Arms: EGO 9mg; Nicotine Free; One High 2,4% nicotine; Own Brand cigarette
Other: nicotine free — smoke, 15 puff, of electronic cigarette nicotine free
  Other Names: categoria electronic cigarette nicotine free "mint".
  Arms: EGO 9mg; One High 2,4% nicotine; Original 7,4 mg nicotine; Own Brand cigarette
Other: Ego 9mg — smoke, 15 puff, of electronic cigarette Ego 9 mg
  Other Names: electronic cigarette Ego 9 mg nicotine
  Arms: Nicotine Free; One High 2,4% nicotine; Own Brand cigarette

SUMMARY:
The aim of the present study is to compare cognitive scores (attention, executive function and working memory) of different e-Cigarette strength with usual cigarettes.

DETAILED DESCRIPTION:
The study is randomised cross-over trial designed to compare: 1) Cognitive performances levels for four different e-Cigarette strength. Participants will be requested to abstain from smoking and alcohol from 20:00 on the night before each study day and from food and caffeine for at least 1 h before the session. On arrival at the study centre, carbon monoxide (CO) will be measured in participants' expired breath. If CO will be >15 parts per million (ppm), the assigned study treatment will be allocated; however, if CO was >15 ppm or they will report smoking in the previous 12 h, participants will be rescheduled wherever possible to a subsequent session.

On the first study day, participants will be randomised to use one of five ordered conditions: Electronic Nicotine Delivery Device (ENDD) (fourth generation) containing nicotine 2,4%; Electronic Nicotine Delivery Device (ENDD (second generation) containing nicotine 7,4 mg; Electronic Nicotine Delivery Device (ENDD containing nicotine 9 mg; Electronic Nicotine Delivery Device (ENDD nicotine free; their usual cigarette. Additionally participants will be trained to use an electronic cigarette. The following tests will be completed at the each visits: Continuous Performance Test - AX version (CPT-AX), Wisconsin card sorting test( WCST), Working memory test (N-BACK).

ELIGIBILITY:
Inclusion Criteria:

* 20 regular smokers (smoking ≥ 15 factory-made cigarettes per day for at least the past 10 years and not currently attempting to quit smoking or wishing to do so in the next 30 days, CO > 10 parts per million ) will be recruited from the local Hospital staff in Catania, Italy.

Exclusion Criteria:

* people who reported recent myocardial infarction, angina pectoris or other serious medical conditions (diabetes mellitus, severe allergies, poorly controlled asthma or other airways disease, poorly controlled psychiatric disorders or current chemical dependence other than nicotine) and
* pregnancy,
* breastfeeding,
* blood pressure > 180 mm Hg systolic and/or 100 mm Hg diastolic,
* weight < 45 or > 120 kg, or
* current use of any other smoking cessation medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-09; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Cognitive Performances | 35 minutes
  Compare cognitive performances in subjects who smoke "Categoria" electronic cigarettes labelled Original 7,4 mg nicotine , "Categoria" electronic cigarettes labelled One 2,4% nicotine, "Categoria" electronic cigarettes labelled "Mint" nicotine free, electronic cigarettes labelled Ego 9 mg nicotine with usual cigarettes.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro per la Prevenzione e Cura del Tabagimso, Catania, Italy, Italy

REFERENCES:
- [Derived] Caponnetto P, Maglia M, Cannella MC, Inguscio L, Buonocore M, Scoglio C, Polosa R, Vinci V. Impact of Different e-Cigarette Generation and Models on Cognitive Performances, Craving and Gesture: A Randomized Cross-Over Trial (CogEcig). Front Psychol. 2017 Mar 9;8:127. doi: 10.3389/fpsyg.2017.00127. eCollection 2017. PMID 28337155